CLINICAL TRIAL: NCT05352932
Title: Establishment of Clinical Staging of Chronic Pancreatitis Based on Histopathology of Pancreatic Duct Biopsy: a Cross-sectional Clinical Study
Brief Title: Establishment of Clinical Staging of Chronic Pancreatitis Based on Histopathology of Pancreatic Duct Biopsy
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Professor, Changhai Hospital
Other Study IDs: ECHO20220321
Record Dates: First submitted 2022-04-24; First posted 2022-04-29 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Chronic Pancreatitis
Keywords: Endoscopic Retrograde Cholangiopancreatography; Histology
MeSH Terms: conditions — Pancreatitis, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Biopsies will be done under ERCP. During the process, biopsy forceps will be used to take one piece of tissue from the wall of the main pancreatic duct in the head and the body of the pancreas. The maximum diameter of each piece of tissue is not less than 1 mm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient group: Patients with chronic pancreatitis or idiopathic recurrent acute pancreatitis are considered as study subjects.
  Interventions: Diagnostic Test: pancreatic duct biopsy

INTERVENTIONS:
Diagnostic Test: pancreatic duct biopsy — Enrolled patients will undergo a baseline assessment, including CP history, clinical symptoms, imaging tests, laboratory tests, etc.
  Then, according to the clinical standard of diagnosis and treatment of chronic pancreatitis, ERCP (with or without Extracorporeal Shock Wave Lithotripsy (ESWL) / endoscopic lithotripsy) will be performed for patients with calculi; pancreatic stent or nasopancreatic stent will be placed for patients with pancreatic duct stenosis. During ERCP, the patient's pancreatic tissue will be biopsied and sent for pathological examination.

SUMMARY:
This study intends to establish the clinical staging of chronic pancreatitis based on histopathology through pancreatic duct biopsy technology.

DETAILED DESCRIPTION:
Chronic pancreatitis (CP) is an inflammatory disease that can causes progressive fibrosis of pancreatic tissue and eventually leads to damage of pancreatic exocrine and endocrine. According to statistics, the prevalence of CP in China is 13/10 million, which is still increasing. Pancreatic duct stones are the most important pathological changes of CP. More than 50% of patients with CP are accompanied by pancreatic duct stones, which can lead to pancreatic duct obstruction, hypertension and tissue ischemia. Removal of pancreatic duct stones under Endoscopic retrograde cholangiopancreatography (ERCP) are the first choice.

Pathological features of CP include pancreatic parenchymal atrophy and interstitial fibrosis resulting from chronic inflammatory damage. Although there are numerous criteria for clinical staging and severity grading of CP, they all have their own limitations, and none of them have been validated by randomized controlled trials. There is also no clear definition of the clinical stage and severity of CP in the guidelines for the diagnosis and treatment of CP. According to the "Clinical Guideline: Chronic Pancreatitis" issued by the American College of Gastroenterology in 2020, histopathology is the "gold standard" for the diagnosis of CP.

In the past ten years, the technology of mother-daughter scope has developed rapidly. The duodenoscope is used as the mother scope, and the cholangiopancreatoscope is used as the daughter scope. The optical fiber or digital imaging system carried by the daughter scope can directly observe the internal situation of the pancreatic and bile ducts. The channel allows the endoscopist to precisely biopsy the wall of the main pancreatic duct with a biopsy forceps. This technology improves the predicament of pancreatic tissue biopsy in the past, allowing ERCP treatment in patients with CP and pancreatic tissue biopsy to be carried out simultaneously.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic pancreatitis or idiopathic recurrent acute pancreatitis;
* In line with the indications for ERCP treatment.

Exclusion Criteria:

* suspected to have malignant tumors;
* history of pancreatic surgery or gastrojejunostomy (Billroth II);
* bile duct stricture secondary to cholangitis or chronic pancreatitis;
* acute pancreatitis exacerbation or acute exacerbation of chronic pancreatitis;
* coagulation dysfunction (INR≥1.5 or platelet count≤50×10^9/L);
* pregnant or breastfeeding women;
* patients who refused to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients meeting the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-03-09 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Histopathological scoring of pancreatic duct biopsy specimens | 14 days after ERCP procedure
  Histopathological evaluations of pancreatic duct biopsies include the presence of ductal squamous metaplasia, the presence of ductal intestinal metaplasia, the presence of ductal dysplasia, the presence of acinar parenchyma, the presence of lobular ducts, the degree of inflammatory cell infiltration (lymphocytes, plasma cells and mast cells) ) and the degree of interstitial fibrosis.

SECONDARY OUTCOMES:
post-ERCP complications | 30 days after ERCP procedure
  Major post-ERCP complications includes post-ERCP pancreatitis, bleeding, infection, and perforation, which are classified as mild, moderate, or severe, depending mainly on the length of hospitalization and the need for invasive treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Liang-hao Hu, MD, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hao L, Liu Y, Xie T, Wang T, Guo HL, Pan J, Wang D, Bi YW, Ji JT, Xin L, Du TT, Lin JH, Zhang D, Zeng XP, Zou WB, Chen H, Li BR, Liao Z, Cong ZJ, Shi RH, Li ZS, Hu LH. Risk Factors and Nomogram for Pancreatic Stone Formation in Chronic Pancreatitis over a Long-Term Course: A Cohort of 2,153 Patients. Digestion. 2020;101(4):473-483. doi: 10.1159/000500941. Epub 2019 Jun 25. PMID 31238312